CLINICAL TRIAL: NCT06413082
Title: Pharmacogenetics of Hypertension: a Single-centre Randomized Study in Patients With Essential Hypertension Treated With Spironolactone or Torasemide
Brief Title: Pharmacogenetics of Torasemide and Spironolactone in Hypertension Treatment
Acronym: ALTUM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Chiara Lanzani, medical doctor in nephrology unit, nephrologist, Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALTUM
Record Dates: First submitted 2023-09-04; First posted 2024-05-14 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Hypertension; Genetic Predisposition; Drug Effect
Keywords: hypertension; genetics; torasemide; spironolactone; pharmacogenetics
MeSH Terms: conditions — Hypertension; Genetic Predisposition to Disease | interventions — Torsemide; Spironolactone; Canrenoic Acid

STUDY DESIGN:
Intervention Model Description: single-center, nationwide, randomized, phase III prospective interventional outpatient study, in two arms, in parallel groups
Who Masked: Participant, Investigator
Masking Description: The study will be double-blind with respect to the genetic analysis and open-label with an observer blind with respect to the primary endpoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Torasemide (Experimental): The study involves the administration of Torasemide 2.5 mg.
  Interventions: Drug: Torasemide
- Spironolactone (Experimental): The study involves the administration of Spironolactone 50 mg orally every day.
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Torasemide — The assignment to each drug will be carried out randomly in each genotypic group with the aim of reaching the same number of patients treated with the two drugs in the different genotypic groups
  Other Names: Demadex; Tortas; Wator; Torsemide
  Arms: Torasemide
Drug: Spironolactone — The assignment to each drug will be carried out randomly in each genotypic group with the aim of reaching the same number of patients treated with the two drugs in the different genotypic groups
  Other Names: Aldactone; Carospir
  Arms: Spironolactone

SUMMARY:
Phase III interventional study to evaluate the different efficacy of Torasemide and Spironolactone in reducing systolic blood pressure in carriers and non-carriers of the different genotypic combinations for Lanosterol and Uromodulin

DETAILED DESCRIPTION:
The investigators will enroll 144 naïve hypertensive subjects who will undertake 2-4 weeks of run-in and 4 weeks of treatment (7 day window at each visit). During this period partecipants will follow a low sodium diet (about 5g/day) and will be monitored with blood chemistry tests

ELIGIBILITY:
Inclusion Criteria:

* male (25-65 years) and female (45-65 years in menopause defined as "12 consecutive months of amenorrhea for which no other physiological or pathological cause has been identified in woman over 45 years of age")
* newly diagnosed hypertensive patients never treated before or on single antihypertensive drug therapy
* hypertension grade I or II (according to 2013 ESH guidelines, in the patient untreated or despite therapy), defined as the following:

  * at visits T-4 and T-2 (week -4 and week -2 ± 7 days, run-in period) the mean of the last 3 consecutive SBP measurements must be >=140 mmHg and/or diastolic BP>= 90mmHg
  * at the T0 visit (week 0 ± 7 days, enrollment), the mean of the last 3 consecutive systolic BP measurements must be >=140 mmHg and <180 mmHg and diastolic BP must be >=90 mmHg and <110 mmHg
* signing of the informed consent for participation in the study and for genotyping.

Exclusion Criteria:

* known causes of secondary hypertension
* stage II hypertension (SBP>= 180 and SBP>=110 mmHg
* history of renal artery stenosis
* significant kidney disease (eGFR-CK-EPI less than 60 mL/min)
* refractory hypokalemia or hyponatremia (Napl < 126 mEq/L)
* hyperkalemia (K > 5.5 mEq/l)
* hypercalcemia
* symptomatic hyperuricemia
* liver disease (transaminases greater than 3 times the maximum laboratory value)
* cardiac pathologies (previous myocardial infarction, atrial fibrillation in progress, etc.)
* diabetes (fasting blood sugar >126mg/dL)

  -. current statin treatment
* obesity (BMI >30 kg/m2)
* ongoing pregnancy
* breastfeeding in progress
* anuria
* hypovolemia and dehydration
* known hypersensitivity to the study drugs (Spironolactone or Torasemide) or to any of the excipients
* ongoing therapy with aminoglycosides or cephalosporins
* participation in a clinical study in which an investigational drug was administered within 30 days or 5 half-lives prior to the study drug
* patients unable to express valid consent

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-09-03 (Actual)

PRIMARY OUTCOMES:
difference in the change of systolic blood pressure(deltaSBP) | week 4 vs. week 0
  the difference in the reduction of systolic blood pressure (deltaSBP) values in essential hypertensive patients who are carriers and noncarriers of the different genotypic combinations for the LSS (lanosterol synthase) and UMOD (uromodulin) genes in response to Spironolactone or Torasemide

SECONDARY OUTCOMES:
difference in diastolic blood pressure change after treatment with Spironolactone or difference in diastolic blood pressure reduction (deltaDBP) | week 4 vs. week 0
  the difference in the reduction of diastolic blood pressure (deltaDBP) values in essential hypertensive patients who are carriers and noncarriers of the different genotypic combinations for the LSS (lanosterol synthase) and UMOD (uromodulin) genes in response to Spironolactone or Torasemide
variation of plasma aldosterone | week 4 vs. week 0
  variation of plasma aldosterone levels in the different genotypic and treatment groups after 4 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Manunta, MD, Study Director — San Raffaele Hospital Milan, Italy
Locations (2):
- Italy (2):
  - San Raffaele Hospital, Milan, Lombardy
  - IRCCS Ospedale San Raffaele, Milan

IPD SHARING:
Plan to Share IPD: No
IDP will be stored in the institutional repository.